CLINICAL TRIAL: NCT04481464
Title: Evaluation of the Efficacy of Chinese Herbal Medicine in Patients With Obesity: a Retrospective Study
Brief Title: Evaluation of the Efficacy of Chinese Herbal Medicine in Patients With Obesity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Shan-Yu Su, Attending Physician, Traditional Chinese Medicine Obstetrics and Gynecology, China Medical University Hospital
Other Study IDs: CMUH109-REC2-101
Record Dates: First submitted 2020-07-15; First posted 2020-07-22 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Obesity
Keywords: obesity; Chinese herbal medicine; efficacy; side effect
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity is defined as abnormal or excessive fat accumulation. It is a complex disease with multifactorial etiology. Although the prevalence of obesity is generally greater in elders and women, obesity rates have increased in all ages and both sexes in recent years. Obesity or overweight also has a higher risk of diabetes, metabolic syndrome, dyslipidemia, hypertension, hyperuricemia, gout, osteoarthritis, cardiovascular disease, coronary artery disease, breast cancer, endometrial cancer and colorectal cancer. The body mass index (BMI), calculated as weight in kilograms divided by the square of height in meters, is widely used to define overweight and obesity in clinical studies. In Taiwan, subjects with BMI between 24 and 27 were diagnosed of overweight, and those with BMI over 27 were diagnosed of obesity.

Chinese herbal medicine (CHM) was widely used in the treatment of obesity. The main purpose of CHM treatment is to promote metabolism, suppress appetite and block intestinal digestion and absorption of fat. Since there are various adverse effects of anti-obesity medicines, and there are surgical complications including infection and anastomotic stenosis, patients may seek CHM for losing weight. Many studies have indicated the efficacy of single herb in the treatment of obesity.

Currently, the amount of computerized clinical data is increasing rapidly with the adoption of electronic medical records. The study is expected to collect the medical records, including the data of body weight, related side effects and biochemical data of each individual. By comparing the change of related data before and after CHM treatment, we could evaluate the efficacy of CHM in patients with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of obesity (ICD-9: 278.00) and received Chinese herbal treatment for obesity in outpatient clinic during January 1, 2007 and December 31, 2019.

Exclusion Criteria:

* Patients who were pregnant or breast feeding during treatment period.
* Patients who were diagnosed of hopothyroidism or Cushing's disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged above 20 years old, diagnosed of obesity (ICD-9: 278.00) and received herbal treatment during january 1, 2007 and December 31, 2019.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Body weight change | The change of body weight is measured monthly from the beginning of the herbal treatment through study completion, an average of 2 years.
  Record the body weight change form the clinical records of obese patients

SECONDARY OUTCOMES:
Side effects | The frequency of side effects is recorded from the beginning of the herbal treatment through study completion, an average of 2 years.
  Record the frequency of side effects from the clinical records of obese patients
Comorbidity | The frequency of comorbidities is recorded from the beginning of the herbal treatment through study completion, an average of 2 years.
  Record the frequency of comorbidities from the clinical records of obese patients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pi-Sunyer X. The medical risks of obesity. Postgrad Med. 2009 Nov;121(6):21-33. doi: 10.3810/pgm.2009.11.2074. PMID 19940414
- [Background] Sun NN, Wu TY, Chau CF. Natural Dietary and Herbal Products in Anti-Obesity Treatment. Molecules. 2016 Oct 11;21(10):1351. doi: 10.3390/molecules21101351. PMID 27727194
- [Background] Cheung BM, Cheung TT, Samaranayake NR. Safety of antiobesity drugs. Ther Adv Drug Saf. 2013 Aug;4(4):171-81. doi: 10.1177/2042098613489721. PMID 25114779
- [Background] Monkhouse SJ, Morgan JD, Norton SA. Complications of bariatric surgery: presentation and emergency management--a review. Ann R Coll Surg Engl. 2009 May;91(4):280-6. doi: 10.1308/003588409X392072. Epub 2009 Apr 2. PMID 19344551
- [Background] Zhang WL, Zhu L, Jiang JG. Active ingredients from natural botanicals in the treatment of obesity. Obes Rev. 2014 Dec;15(12):957-67. doi: 10.1111/obr.12228. Epub 2014 Nov 23. PMID 25417736
- [Background] Choi JS, Kim JH, Ali MY, Min BS, Kim GD, Jung HA. Coptis chinensis alkaloids exert anti-adipogenic activity on 3T3-L1 adipocytes by downregulating C/EBP-alpha and PPAR-gamma. Fitoterapia. 2014 Oct;98:199-208. doi: 10.1016/j.fitote.2014.08.006. Epub 2014 Aug 12. PMID 25128422
- [Background] Kho MC, Lee YJ, Park JH, Kim HY, Yoon JJ, Ahn YM, Tan R, Park MC, Cha JD, Choi KM, Kang DG, Lee HS. Fermented Red Ginseng Potentiates Improvement of Metabolic Dysfunction in Metabolic Syndrome Rat Models. Nutrients. 2016 Jun 16;8(6):369. doi: 10.3390/nu8060369. PMID 27322312
- [Background] Karu N, Reifen R, Kerem Z. Weight gain reduction in mice fed Panax ginseng saponin, a pancreatic lipase inhibitor. J Agric Food Chem. 2007 Apr 18;55(8):2824-8. doi: 10.1021/jf0628025. Epub 2007 Mar 17. PMID 17367157
- [Background] Kim BS, Song MY, Kim H. The anti-obesity effect of Ephedra sinica through modulation of gut microbiota in obese Korean women. J Ethnopharmacol. 2014 Mar 28;152(3):532-9. doi: 10.1016/j.jep.2014.01.038. Epub 2014 Feb 17. PMID 24556223
- [Background] Li J, Ding L, Song B, Xiao X, Qi M, Yang Q, Yang Q, Tang X, Wang Z, Yang L. Emodin improves lipid and glucose metabolism in high fat diet-induced obese mice through regulating SREBP pathway. Eur J Pharmacol. 2016 Jan 5;770:99-109. doi: 10.1016/j.ejphar.2015.11.045. Epub 2015 Nov 25. PMID 26626587
- [Background] Liu Y, Sun M, Yao H, Liu Y, Gao R. Herbal Medicine for the Treatment of Obesity: An Overview of Scientific Evidence from 2007 to 2017. Evid Based Complement Alternat Med. 2017;2017:8943059. doi: 10.1155/2017/8943059. Epub 2017 Sep 25. PMID 29234439